CLINICAL TRIAL: NCT04749303
Title: Impact of Screen Size on Colorectal Adenoma Detection Rate: a Single Centre Randomised Controlled Trial
Brief Title: Impact of Screen Size on Colorectal Adenoma Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Tony Wing Chung Mak, Clinical Associate Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020.327
Record Dates: First submitted 2021-02-02; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Colon Polyp; Colon Adenoma; Colorectal Neoplasms
Keywords: Colonoscopy; Adenoma Detection Rate; Colorectal cancer screening; Screen size
MeSH Terms: conditions — Colonic Polyps; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Large screen vs standard screen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large screen (Active Comparator): This is a high definition screen which gives a 76cm height and 67cm width (area: 5092cm2) endoscopic image.
  Interventions: Procedure: Large Screen
- Standard screen (No Intervention): This is a high definition screen which gives a 37.5cm height and 32.5cm width (area: 1218.75cm2) endoscopic image.

INTERVENTIONS:
Procedure: Large Screen — Large screen size is 4x larger than standard screen, we hope that the colonoscopies carried out with large screens will confer to better lesion detection
  Other Names: Standard Screen
  Arms: Large screen

SUMMARY:
The purpose of this study is to assess whether the use of large screen during colonoscopy will increase adenoma detection rate.

DETAILED DESCRIPTION:
Colorectal cancer is the 3rd most common cancer in the world. Recently in Hong Kong it has surpassed lung cancer to be the most common cancer. Hence it is essential not only to have up-to-date surgical and oncological treatment but also a need an effective preventative strategy.

In the past few decades, removal of pre-malignant colonic lesions such as adenomas have been shown to prevent development of colorectal cancers. Colonoscopy is currently the only technique which can perform both detection and treatment during the same procedure. However, concerns have been raised about the effectiveness of colonoscopy in the prevention of CRC after several studies reported unexpected high incidence rates of interval carcinomas (IC), especially in the proximal colon. Most ICs are suspected to arise from missed colon lesions during colonoscopy. Factors concerning missed colonic lesions are multifactorial such as adequate bowel preparation, skill level of endoscopists, the number of endoscopy staff in the room as "eyes" to help with polyp detection and withdrawal time.

Following a pilot study in our endoscopy unit, we believe the size of the screen projecting the endoscopic image may have a positive influence on adenoma detection. Therefore, we feel that a well-designed and adequately powered randomised controlled trial may help to confirm this.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above
* Referred to the endoscopy unit for diagnostic or surveillance colonoscopy

Exclusion Criteria:

* Familial history of Familial adenomatous polyposis or Hereditary non-polyposis colorectal cancer
* Known history of inflammatory bowel disease
* Emergency endoscopy of any nature (such as for gastrointestinal bleeding, assessment of large bowel investigation and colonic decompression)
* Patients with colostomy
* Previously incomplete colonoscopy (not including insufficient preparation)
* Patients with known palliative colorectal malignant disease Patients with coagulopathies Inability to give informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 656 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Adenoma Detection Rate (ADR) | 12 months
  ADR is defined as the proportion of an endoscopist's screening colonoscopies in which one or more adenomas have been detected in patients

SECONDARY OUTCOMES:
Mean number of adenomas detected per colonoscopy | 12 months
  Mean number of adenomas detected per colonoscopy found in each arm
Mean number of sessile serrated polyps | 12 months
  Mean number of sessile serrated polyps found in each arm
Caecal intubation rate | 12 months
  percentage of caecal intubation rate in each arm
Bowel cleansing level | 12 months
  According to the Boston bowel preparation scale (0=worst bowel preparation to 9= best bowel preparation). Comparison of each arm.
Procedure Time | 12 months
  Both intubation and withdrawal time will be recorded. Comparison of each arm.
Severe adverse events | 12 months
  SAEs of both arms for comparisons

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No